CLINICAL TRIAL: NCT01330108
Title: Safely Change From Bosentan to Ambrisentan in Pulmonary Hypertension
Acronym: SCOBA-PH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOBA-PH
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; WHO Group 1
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ambrisentan (Experimental): patients currently on bosentan to ambrisentan for the treatment of pulmonary arterial hypertension.
  Interventions: Drug: ambrisentan

INTERVENTIONS:
Drug: ambrisentan — ambrisentan 2.5mg, 5mg, & 10mg. Daily dosage.
  Other Names: Letairis

SUMMARY:
The primary objective of this study is to assess the safety and tolerance of changing patients currently on bosentan to ambrisentan for the treatment of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
The therapy of pulmonary arterial hypertension (PAH) has been revolutionized with the development and subsequent instruction of oral endothelin receptor antagonists (ERA). The first approved ERA, bosentan (Tracleer, Actelion, Inc.) is an effective drug widely used throughout the world in the therapy of PAH. Newer ERA's, with purported advantages over the first approved drug have since been tested and subsequently been approved for the therapy of PAH in the USA and other countries including ambrisentan (Letairis, Gilead Sciences, Inc.). However, there is little data available on the efficacy, safety and tolerability of the elective change from oral bosentan to oral ambrisentan in PAH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients followed routinely in the pulmonary vascular disease clinic at the University of Alabama in Birmingham, greater than or equal to 19 years of age.
2. World Health Organization (WHO) PAH Type I
3. WHO class I-IV symptoms (no functional class exclusion).
4. On bosentan, twice a day, with a maximum daily dose of 250mg, on a stable dose for 3 months with no clinical indication to discontinue the drug (i.e., increased liver function studies or other intolerance). Patients may be on other drug therapies for PAH, and also may be on oxygen therapy (intermittent or continuous).

Exclusion Criteria:

1. Known intolerance or allergy to ambrisentan.
2. Prior therapy with ambrisentan.
3. Current therapy with two phosphodiesterase-5 inhibitors.
4. Change in other approved therapy for PAH (including phosphodiesterase-5 inhibitors and prostanoids) within 4 weeks of baseline study visit.
5. Planned addition of prostanoid for clinical reasons within 3 months of baseline study visit.
6. Active participation in another clinical study involving the medical therapy of PAH.
7. Uncontrolled systemic hypertension or angina pectoris
8. Serum creatinine greater than 2.5 at or within 4 weeks of baseline.
9. Serum liver function studies greater than 3 x normal at or within 4 weeks of baseline study visit.
10. In the opinion of the investigator, a change in PAH therapy would present significant risk to the subject.
11. In the opinion of the investigator, the participant is unlikely to survive for 12 weeks after study entry.
12. In the opinion of the investigator, the participant is likely to undergo lung or heart-lung transplantation within 12 weeks of study entry.
13. A woman of childbearing potential who is not using an acceptable form of contraception.
14. Pregnancy.
15. In the opinion of the investigator, a participant who is not capable or willing to follow the study procedures.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Bourge, MD, Principal Investigator — Univerisity of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ambrisentan
Started | 32
Completed | 28
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Subjects described in baseline are those that completed the study
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Not Able to Tolerate Ambrisentan
Description: If a subject was not able tolerate ambrisentan, subject was returned to use of bosentan and ambrisentan was withdrawn within first 12 weeks of start. A subject was considered to not be able to tolerate ambrisentan if they experienced an adverse event or side effect that was not acceptable to the subject.
Time Frame: baseline to 12 weeks
Measure: Number; unit: participants
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
participants | 4

2. Secondary Outcome: Mean Change in Distance for a Six Minute Walk at 12 Weeks Post Start of Ambrisentan
Description: Evaluate the change in exercise tolerance. Measured the distance a subject was capable of walking in 6 minutes at basline compared to the distance at 12 weeks. The distance was measured in meters. A postive result reflects the distance increased at 12 weeks, a negative result reflects how much shorter the distance was.
Time Frame: baseline to 12 weeks
Measure: Mean (Full Range); unit: meters
Arm/Group | Ambrisentan
Number analyzed (Participants) | 28
meters | 368.71 [190 to 510]

ADVERSE EVENTS:
Arm/Group | Ambrisentan
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan (N=32)
edema (Cardiac disorders) | 10 (10)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
rash, not attibuted to drug (Skin and subcutaneous tissue disorders) | 1 (1)
lower extremity edema (Cardiac disorders) | 2 (2) — resolved post withdrawl of drug

LIMITATIONS AND CAVEATS:
There is bias in the study due to the fact that subjects have been proven to tolerate the initial drug in the study (bosentan) and adequate time was not allowed for subjects to be able to tolerate ambisentan

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No